CLINICAL TRIAL: NCT04851132
Title: Radiotherapy Plus Durvalumab in Elderly Esophageal Squamous Cell Carcinoma: A Prospective Phase II Clinical Trial
Brief Title: Radiotherapy Plus Durvalumab in Elderly Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhouguang Hui, M.D., Chief physician, Director of VIP Department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2840
Record Dates: First submitted 2021-04-05; First posted 2021-04-20 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy; durvalumab

STUDY DESIGN:
Intervention Model Description: RT + Durvalumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exprimental Arm (Experimental): IMRT plus Durvalumab
  Interventions: Radiation: Radiotherapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Radiotherapy — IMRT (Intensity Modulated RT) or 3D-CRT (three-dimensional conformal radiotherapy); 95% PGTV 59.92Gy/2.14Gy/28f; 95% GTVnd 59.92Gy/2.14Gy/28f; 95% PTV 50.40Gy/1.80Gy/28f; 5 days a week; 6 weeks.
Drug: Durvalumab — Durvalumab 1000 mg, intravenously (IV), on Day 1 of radiotherapy, every 3 weeks for up to 18 administrations.

SUMMARY:
The incidence and mortality of esophageal cancer are at the forefront in China, among which the elderly patients account for a large proportion. Concurrent chemoradiotherapy is the standard treatment for inoperable locally advanced esophageal cancer. Most elderly patients with esophageal cancer cannot tolerate concurrent chemotherapy because of complications and other reasons. Immunotherapy has definite efficacy and low toxicity in advanced esophageal squamous cell carcinoma, and the results combined with radiotherapy have also been preliminarily reported. Therefore, it is necessary to further explore the efficacy and safety of radiotherapy combined with immunotherapy in elderly patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 70-85 years old, both men and women
2. Histologically confirmed esophageal squamous cell carcinoma located in thoracic segment, treatment naive
3. Stage cT2-4aNanyM0 (AJCC 8 TNM classification)
4. Unresectable, unable to tolerate or refuse surgery and concurrent chemoradiotherapy
5. ECOG PS 0-2
6. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
7. No severe abnormalities of the Hematologic system, heart, lung, liver, kidney, and immunodeficiency
8. Adequate bone marrow and organ function as defined below (excluding the use of any blood components and cell growth factors within 7 days):

   * Absolute neutrophil count≥1,500/mm3
   * Platelets ≥ 100,000/mm3
   * Hemoglobin ≥ 5.6 mmol/L (9g/dL)
   * Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥50 mL/min by Cockcroft-Gault estimation
   * Total bilirubin ≤ 1.5 x ULN
   * ALT and AST ≤ 2.5 x ULN
   * Proteinuria < 2+, for subjects with urine protein ≥ 2 + at baseline, urine samples should be collected within 24 hours and urine protein in 24 hours should be ≤ 1g
9. INR or PT or aPTT ≤ 1.5 x ULN
10. Life expectancy more than 6 months
11. Ability to understand and willingness to sign an IRB approved written informed consent document, and capable of proper therapeutic compliance, and accessible to correct follow-up

Exclusion Criteria:

1. Complete esophageal obstruction that unable to eat fluid and cannot provide necessary nutrition through nasal feeding
2. Patients with obvious ulcer or esophageal perforation or hematemesis
3. Placement of esophagotracheal stents
4. Has a history or current evidence of pulmonary fibrosis, interstitial pneumonia, pneumonoconiosis, drug-associated pneumonia, severe impairment of pulmonary function
5. Has had major surgery within 28 days prior to the start of the treatment
6. Immunosuppressive drugs used within 4 weeks prior to the initial study treatment, excluding local glucocorticoids, or systemic glucocorticoids at physiological doses (i.e., no more than 10 mg/ day of prednisone or equivalent doses of other glucocorticoids);
7. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, glomerulonephritis, thyroiditis (patients with vitiligo or asthma has been completely relieved in childhood, and do not need any intervention during adulthood can be included; patients with type I diabetes with good insulin control can also be included; hypothyroidism caused by autoimmune thyroiditis requiring hormone replacement therapy can also be included)
8. Has had congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV-DNA ≥ 104 copies/ml) or hepatitis C (HCV-RNA ≥ 103 copies/ml; For chronic hepatitis B virus carriers, HBV viral load must be < 2000 IU/ml (< 104 copies / ml), and must receive antiviral therapy at the same time before they can be enrolled
9. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
10. Uncontrolled clinically significant disease, including active infection, uncontrolled hypertension, unstable angina pectoris, angina within the past 3 months, heart failure > NYHA II, myocardial infarction within the past 6 months, severe arrhythmias requirement for treatment or intervention, liver/kidney or metabolic disease
11. System infections that require treatment
12. Received a live vaccine within 4 weeks of the first dose of study medication
13. Synchronous or metachronous second primary malignancy. Participants with basal cell carcinoma of the skin, or cervical cancer in situ that have undergone potentially curative therapy are not excluded from the study
14. Patients who have participated in other clinical trials within 30 days
15. Drug addiction, chronic alcoholism and AIDS
16. Patients with uncontrollable seizures or loss of self-control due to mental illness
17. Those with a history of severe allergy or specific physique
18. The investigators judge not suitable for inclusion

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1-year
  PFS was assessed by Response Evaluation Criteria in Solid Tumors (RECIST)1.1. Progression-free survival defined as the time from enrollment to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 1-, 2- and 3-year
  Overall survival defined as the time from enrollment to death due to any cause.
Progression-free survival (PFS) | 2- and 3-year
  PFS was assessed by Response Evaluation Criteria in Solid Tumors (RECIST)1.1. Progression-free survival defined as the time from enrollment to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.
Objective Response Rate (ORR) | during the intervention up to 60 weeks
  ORR was Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Disease Control Rate (DCR) | during the intervention up to 60 weeks
  DCR was Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Number of participants with an adverse event | Up to 60 weeks
  Evaluanted by CTCAE 5.0
Quality of Life (QOL): questionnaire EORTC QLQ-C30 (version 3) | up to 60 weeks
  Evaluate the quality of life via questionnaire EORTC QLQ-C30 (version 3), minimum value 30, maximum value 126, higher scores mean a worse outcome.

OTHER OUTCOMES:
Quality of Life (QOL): questionnaire EORTC QLQ-OES18 | up to 60 weeks
  Evaluate the quality of life via questionnaire EORTC QLQ-OES18, minimum value 18, maximum value 72, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No